CLINICAL TRIAL: NCT06078943
Title: ABL90 Flex Plus Method Comparison Neonatal Arterial, Venous, Capillary Blood
Brief Title: ABL90 FP MC Neonatal Arterial, Venous, Capillary Blood
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radiometer Medical ApS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: DC-083185
Record Dates: First submitted 2023-02-14; First posted 2023-10-12 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-01

CONDITIONS: Congenital Heart Disease
Keywords: Blood gas
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Investigational Device (Active Comparator): The test device in this clinical study is the ABL90 FLEX PLUS running SW3.5 MR2 manufactured by Radiometer Medical ApS The analyzer provides results for 17 parameters in 35 seconds using 65 µL heparinized whole blood. However, in this investigation only the data concerning the parameters ctBil and FHbF will be evaluated.
  Interventions: Device: method comparison
- Predicate device (Sham Comparator): The predicate device for this study is the unmodified device ABL90 FLEX PLUS (k160153) running software SW 3.1 MR7 including sensor casettes and solution packs versions corresponding to 2016.
  ABL90 FLEX PLUS SW 3.1 MR7, has been selected as the predicate device because it has the appropriate 510(k) clearance, and the intended use matches the ABL90 FLEX PLUS SW. SW3.5 MR2 device.
  Interventions: Device: method comparison

INTERVENTIONS:
Device: method comparison — to quantify the relationship using comparison measurement from the same sample between ABL90 FLEX PLUS and the predicate device within the reportable range for all ctBil and FHbF in heparinized arterial and venous neonatal whole blood in syringe measuring mode (S65, SP65) and heparinized mixed venous/arterial whole blood samples in capillary measuring mode (C65)

SUMMARY:
The goal of this clinical trial is to validate performance claims for method comparison for ABL90 FLEX PLUS in heparinized neonatal arterial, venous, and capillary whole blood for ctBil and FHbF in a Point of Care (POC) setting.

DETAILED DESCRIPTION:
The main question it aims to answer is:

To quantify the relationship using comparison measurement from the same sample between the test device and the predicate device within the reportable range for ctBil and FHbF in heparinized arterial and venous neonatal whole blood in syringe measuring mode (S65, SP65) and heparinized mixed venous/arterial whole blood samples in capillary measuring mode (C65).

ELIGIBILITY:
Inclusion Criteria:

* The following are the inclusion criteria for the neonatal subjects:

  * The age of the subject must be ≤28 days.
  * Subject evaluated as suitable according to the protocol to enroll in the study by principal investigator or designee.
  * Subjects having a sample drawn as part of standard of care that meets the requirements for samples in this study.

The following are the inclusion criteria for the subjects providing placenta for cord blood:

• Delivery ≥38 weeks of gestation.

Exclusion Criteria:

* The following are the exclusion criteria for the neonatal subjects:

  * Subject who has already provided successful results from arterial, venous and mixed venous/arterial samples, to cover both syringe modes and the capillary mode and parameters.
  * Subjects exposed to the substances listed in Appendix 1 with last dose within 72 hours, should be excluded due to risk of interference.
  * Subjects with known infectious disease such as Hepatitis C and HIV (in order to ensure the operator safety).

The following are the exclusion criteria for the subjects providing placenta for cord blood:

• Subjects positive of HIV or Hepatitis C

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 612 (Estimated)
Dates: Start 2023-03-17 (Actual); Primary Completion 2024-01-13 (Estimated); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
Slope, R^2 and bias | 6-9 months
  Slope, R^2 and bias at medical decision points for each combination of modes and sample type

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Dietzen, PhD, Principal Investigator — St. Louis Children's Hospital
Locations (1):
- St Louis Children's Hospital, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No